CLINICAL TRIAL: NCT03035682
Title: The Impact of a mHealth Application on Outpatient Physical Therapy HEP Adherence and Outcomes: A Randomized Clinical Trial
Brief Title: The Impact of a mHealth Application on Outpatient Physical Therapy HEP Adherence and Outcomes: A RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aultman Health Foundation (Other)
Responsible Party: Principal Investigator, Robert Elson PT, Physical Therapist, Aultman Health Foundation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016.11RE
Record Dates: First submitted 2017-01-18; First posted 2017-01-30 (Estimated); Last update posted 2020-08-25 (Actual); Status verified 2020-08

CONDITIONS: Orthopedic Disorder; Musculoskeletal Injury
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional Group (Active Comparator): The control group will receive traditional PT services as deemed clinically appropriate via examination to include traditional home exercise prescription.
  Interventions: Other: Traditional Group
- Augmented Media Group (Experimental): The Augmented Media group will receive traditional PT services as deemed clinically appropriate via examination and include home exercise prescription via a mobile health application.
  Interventions: Other: Augmented Media Group

INTERVENTIONS:
Other: Augmented Media Group — The intervention group will receive traditional PT services deemed clinically appropriate via examination plus home exercise prescription augmented via a mobile health application. The augmented media group will receive digital exercise prescription via a mobile health application source (Physitrack) that includes: high definition video and pictures, education material and written instruction, reminder notification and in-app logging of completion.
  Arms: Augmented Media Group
Other: Traditional Group — The Traditional Group will receive traditional PT services deemed clinically appropriate via examination plus traditional home exercise prescription.
  Arms: Traditional Group

SUMMARY:
The purpose of this study is to determine the impact a mobile health application has on adherence to a physical therapy home exercise program and its effect on functional outcomes.

DETAILED DESCRIPTION:
Outpatient physical therapy is an integral aspect in combating the impairment and dysfunction associated with musculoskeletal injuries. Healthcare and insurance restrictions are leading to reduced clinic visits, encouraging efficient and effective treatments and focusing a greater demand on education, proactive wellness and home exercise maintenance. Home exercise prescription has long been a fundamental aspect to a physical therapy routine or regimen. It is well established that exercise protocols can positively impact pain, fitness levels, physical function and measures of life quality (Forkan, Pumper, Smyth, Wirkkala, A Ciol, & Shumway-Cook, 2006). It is also recognized that treatment outcomes may be negatively impacted by non-adherence to the prescribed exercise recommendation in rehabilitation (Holden, Haywood, Portia, Gee, & Mclean, 2014). Research historically suggests that levels of non-adherence to exercise prescription range from 50-70% (Bassett, 2003; Sluijs, Kok, & van der Zee, 1993), and likely increase as time passes. Investigating non-adherence demonstrates a myriad of influencing factors. These factors can be characterized as motivators and barriers. With the explosion of mobile communications access and increasing number of active device users, healthcare is embarking on the concept of mobile health management. Mobile health interventions have been found to have a positive impact in the arenas of medication compliance, weight loss, chronic disease management and postoperative complication (Lee, 2016; Ronghua, Li, (2015).The implementation of a mobile health application in physical therapy outpatient management has not been well established. It is time to investigate the impact of using a mobile health application on a prescribed physical therapy treatment regimen for the enhancement of HEP adherence and functional outcome assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Any musculoskeletal pathology: spine, UE, LE
2. Age18 or older
3. Primary language is English. Ability to read, write and understand the English language
4. Ownership of mobile smart phone
5. Functional and cognitive ability to operate/manipulate a mobile media application
6. Willingness to use their data package for support/use of mobile application

Exclusion Criteria:

Following the initial screening criteria, the study population will be scrutinized for exclusion.

Exclusion criteria:

1. History of neurological pathology with neurological impairments
2. Impaired cognition
3. Difficulty with operation and manipulation of mobile application
4. Difficulty with directions as set forth by the intake The exclusion criteria will be screened by written intake and a traditional medical history by the primary researcher. Subject enrollment will commence after eligibility is met and informed consent received.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2017-01-23 (Actual); Primary Completion 2018-07-23 (Actual); Study Completion 2019-12-12 (Actual)

PRIMARY OUTCOMES:
Adherence Exercise Logs: Adherence = exercise reps completed (x) sets completed (x) times per day completed (x) days per week completed divided by total number of (reps) (sets) (time per day) (days per week) assigned to the HEP regimen for each patient | Weekly during course of patient standard treatment. Logs will be assessed over each 7 day period after initial treatment session and collected up to a period of 24 weeks or discharge from therapy intervention for any reason, which ever may occur first.

SECONDARY OUTCOMES:
Self -report Adherence Question: Both groups will complete a single question assessment regarding their perceived level of adherence to the prescribed home exercise plan. | Completed at 1 week after inital exam , at discharge from PT as defined by a period up to 24 weeks or discontinuation of therapy intervention for any reason, which ever may occur first, and 3 month follow-up. 6month follow-up if subject agreeable.
Numeric Pain Rating Scale (NPRS) 0-10 scale. | Outcome will be completed at initial exam, at discharge from PT as defined by a period up to 24 weeks or discontinuation of therapy intervention for any reason, which ever may occur first.
Patient-Specific Functional Scale (PSFS) | Outcome will be completed at initial exam, at discharge from PT as defined by a period up to 24 weeks or discontinuation of therapy intervention for any reason, which ever may occur first.
The Global Rating of Change Scale (GROC) | At patient discharge from PT as defined by a period up to 24 weeks or discontinuation of therapy intervention for any reason, which ever may occur first, and at 3 month follow-up. 6month follow-up if subject agreeable.

CONTACTS AND LOCATIONS:
Overall Officials: Robert A Elson, MPT, Principal Investigator — Aultman Health Foundation
Locations (1):
- Aultman Hospital - West Physical Therapy, Canton, Ohio, United States

IPD SHARING:
Plan to Share IPD: No